CLINICAL TRIAL: NCT05676229
Title: The Use of a Probiotic Blend in Reducing Anthropometric Measurements and Improving Biochemical Parameters in Adults With Overweight and/or Obese
Brief Title: Probiotic Blend in Reducing Anthropometric Measurements in Obese Adults
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Responsible Party: Principal Investigator, Monique Michels, PhD, Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 65117022.1.0000.0119
Record Dates: First submitted 2022-12-09; First posted 2023-01-09 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Obesity; Endocrine; Overweight and Obesity; Overweight, Obesity and Other Hyperalimentation
Keywords: obesity; probiotic; supplement
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Randomised, triple-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Volunteers supplemented with maltodextrin
  Interventions: Dietary Supplement: Placebo
- Probiotic Blend (Active Comparator): Lactobacillus gasseri CCT 7850 and Bifidobacterium lactis CCT 7858 - Final concentration: 1 x 10e10 UFC/ day
  Interventions: Dietary Supplement: Probiotic blend

INTERVENTIONS:
Dietary Supplement: Probiotic blend — Lactobacillus gasseri CCT 7850 and Bifidobacterium lactis CCT 7858
  Arms: Probiotic Blend
Dietary Supplement: Placebo — Maltodextrin only (vehicle)
  Arms: Placebo

SUMMARY:
It is already known that dysbiosis, that is, qualitative and quantitative changes in the composition of the intestinal microbiota, can be associated with the development of a series of intestinal and extra-intestinal disorders. Dysbiosis is reported in irritable bowel syndrome, inflammatory bowel disease, colorectal cancer, allergic diseases, non-alcoholic steatohepatitis, arteriosclerotic diseases, neurological diseases and metabolic syndromes, mainly diabetes and obesity. Among the many factors that play a key role in obesity, a number of studies show the intestinal microbiota as an important contributor. Many studies carried out with probiotics have shown that their administration can be effective in the prevention and treatment of obesity. Furthermore, it is found that benefits for body weight, abdominal adiposity, anthropometric measurements and body composition are often associated with favorable metabolic effects.

DETAILED DESCRIPTION:
Obesity is defined as excessive accumulation of body fat, caused by an energy imbalance. Approximately 13% of the world's adult population is obese, and in Brazil 19.8% of adults are obese. This disease is a risk factor for the development of other non-communicable chronic diseases (NCDs), such as: type 2 diabetes mellitus (DM2), dyslipidemia, cardiovascular diseases, musculoskeletal disorders and some types of cancer. It is a complex and multifactorial disease, which is why it is considered difficult to control and a cause for global concern. Among the causes of the disease, genetic, environmental and psychological factors can be mentioned, in addition to the interference of the intestinal microbiota, among others.

The interaction of the intestinal microbiota with the host has been studied through metabolomics, in order to understand the influence that the microbiota can exert on the functioning of the host organism. The study of the profile of low molecular weight metabolites of biological fluids such as serum/plasma and urine aims to understand the metabolic changes that occur in individuals with obesity, encompassing the understanding of the mechanisms of the disease.

Studies have shown differences in the metabolic profile of obese individuals compared to eutrophic individuals, with a positive correlation between body mass index (BMI) and increased concentrations of chain amino acids (BCAA) and glutamate. The gut microbiota appears to play a crucial role in host metabolism, being a pathway through which it leads to changes associated with obesity.

In this context, the intestinal microbiota can be modulated by prebiotics, probiotics and symbiotics, promoting changes in its composition, resulting in the regeneration of the intestinal barrier and, with that, ceasing metabolic endotoxemia and low-grade inflammation.

In addition, they have effects on the modulation of the immune system, regulating the production of pro and anti-inflammatory cytokines, reducing IR. Through these mechanisms, probiotics and symbiotics alter the microbiota profile of individuals leading to loss of body weight and metabolic parameters associated with obesity.

Several studies have shown beneficial effects of using probiotics on body weight, glycemic control, improvement in lipid profile and blood pressure (BP). However, there are controversies about which are the best strains for this purpose. There are five systematic reviews currently published with or without meta-analysis that address the effect of using different probiotics on body weight. Among the strains associated with weight loss and/or adiposity, L. plantarum associated with L. rhamnosus and hypocaloric diet stand out; L. plantarum with L. curvatus; L. gasseri; L. amylovorus; L. acidophilus and L. casei associated with phenolic compounds; or Lactobacillus mix.

ELIGIBILITY:
Inclusion Criteria:

* Provision of Free and Informed Consent in writing, signed and dated;
* Age according to the indicated population (18-65 years old)
* both genders;
* Body mass index (BMI) of 25 - 35 Kg/m2.

Exclusion Criteria:

* Pregnant and lactating women
* Individuals with a history of daily consumption of probiotics, fermented milk and/or yogurt; subjects known to have demonstrated a prior reaction, including anaphylaxis, to any substance in the composition of the study product;
* Individuals with concomitant participation in another clinical trial;
* History of autoimmune, cardiovascular, thyroid, or chronic liver disease;
* Making use of medication capable of affecting weight change, antidiabetic medication, hypolipidemic agents;
* Individuals who have undergone weight loss surgery,
* Weight change greater than 5% in the last three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-02-19 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Body fat composition by Bioelectrical impedance analysis | three months
  By Bioelectrical impedance analysis (BIA). This is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body.

SECONDARY OUTCOMES:
Total cholesterol by blood analyses | three months
  biochemical analyses before and after inclusion: Total cholesterol to be carried out in a reference laboratory. Total cholesterol will be measured in mg/dL
quality of life questionnaire score | three months
  quality of life and improvement of gastrointestinal symptoms by SF-36 scale (It comprises 36 questions that cover eight domains of health)
Gastrointestinal Symptom Rating Scale (GSRS) questionnaire score | three months
  GSRS scale: An interview-based rating scale consisting of 15 items for assessment of gastrointestinal symptoms
Weight | three months
  weight will be measured in kilograms
height | three months
  height will be measured in centimeters
HDL levels by blood analyses | three months
  biochemical analyses before and after inclusion: HDL to be carried out in a reference laboratory. HDL will be measured in mg/dL
LDL levels by blood analyses | three months
  biochemical analyses before and after inclusion: LDL to be carried out in a reference laboratory. LDL will be measured in mg/dL
triglycerides levels by blood analyses | three months
  biochemical analyses before and after inclusion: triglycerides to be carried out in a reference laboratory. triglycerides will be measured in ml/dL
Glucose levels by blood analyses | three months
  biochemical analyses before and after inclusion: glucose to be carried out in a reference laboratory. glucose will be measured in mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade do Extremo Sul Catarinense, Criciúma, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Undecided